CLINICAL TRIAL: NCT04919876
Title: The Impact of a Phytochemical Supplement on "Metabolic Aging" in Older Overweight Adults Relative to Young Lean Adults
Brief Title: Phytochemicals on "Metabolic Aging" in Older Overweight Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biofortis, Merieux NutriSciences (Industry)
Responsible Party: Principal Investigator, Oliver Chen, Director of Nutrition Science and Biostatistics, Biofortis, Merieux NutriSciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2920
Record Dates: First submitted 2018-04-10; First posted 2021-06-09 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Mitochondrial Functions
Keywords: phytochemicals, fruit, vegetables, older adults
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo-controlled, parallel design, controlled feeding trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: capsules for 2 supplement have the same color and shape
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fruit/vegetable supplement (FVS) (Experimental): The experimental product will be prepared by combing Juice Plus+ Garden Blend, Juice Plus+ Orchard Blend, and Juice Plus+ Berry Blend in an equal proportion.
  Interventions: Dietary Supplement: fruit/vegetable supplement (FVS)
- placebo (Placebo Comparator): The placebo comprises microcrystalline cellulose and 0.5% magnesium stearate.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: fruit/vegetable supplement (FVS) — The supplement contains polyphenols, carotenoids, and other phytochemicals present in plant foods.
  Arms: fruit/vegetable supplement (FVS)
Dietary Supplement: Placebo — The product does not contain nutrients present in the FVS.
  Arms: placebo

SUMMARY:
Aging is a complex and inevitable biological process that is associated with numerous chronic health conditions and the development and progression of diseases. It is manifested partly by a progressive decline in fitness and an increase in death. The key to healthy aging is a healthy lifestyle, including eating a variety of healthy foods and frequently participating in physical activities. Supplements made from widely consumed plant products have the potential for promoting healthy aging. However, more human data is required to substantiate this potential. Thus, the purpose of this study is to determine examining whether older adults taking a fruit/vegetable supplement for 6 weeks will have biochemical values of stool, blood, and urine similar to those of younger adults. The fruit/vegetable supplement contains a variety of vitamins and minerals and other nutrients that have been known to be beneficial to human health and many Americans may consume inadequate amounts in their daily diet. In order for us to understand how these nutrients may benefit health, we are interested in determining whether they can modify biochemical values of blood that occur in the body after taking the supplement for 6 weeks. We aim to have 40 older subjects and 20 younger subjects complete the trial. The enrolled subjects will consume prepackaged study meals for approximately 8 weeks and provide blood samples. The study meals will comprise foods most Americans eat every day. The older subjects, but not younger subjects, will take the assigned supplement. The younger subjects will consume the study meals for 2 weeks and provide one blood sample during the study.

DETAILED DESCRIPTION:
Advanced age is associated with reduced mitochondrial capacity and altered metabolomic signatures relative to those at younger ages. We hypothesize that supplemental fruit and vegetable phytochemicals will slow or reverse signs of metabolic aging by enhancing mitochondrial capacity in older, overweight/obese adults as well as shift their metabolomic signature toward those of younger, leaner adults. To test this hypothesis, we will pursue the following specific aims in a controlled feeding trial to diminish the confounding effect of concurrent and confounding dietary factors.

Specific Aim 1: To determine the extent to which supplemental fruit and vegetable concentrates will shift the mitochondrial capacity of peripheral blood mononuclear cells in older, overweight older adults toward that of young, lean adults.

Specific Aim 2: To determine the extent to which supplemental fruit and vegetable concentrates will shift the plasma metabolomic signature of older, overweight adults toward that of young, lean adults.

The experimental design is a randomized, double-blind, placebo-controlled, parallel design, controlled feeding trial. This trial will enroll 40 older adults, as well as 20 younger adults to serve as a reference, to complete the study. They will be generally healthy. The older adults will be ≥55 y and have BMI >27.0 and <35 kg/m2, and the younger adults will be 18-30 y and have BMI >18.5 and <27 kg/m2. The older subjects will be randomized to receive either placebo (PLA) or fruit/vegetable supplement (FVS) for 6 weeks after a 2-wk run-in period. The younger adults serving as the reference group for the older subjects will only participate in the run-in period and will not receive any dietary supplements. During the whole study, including the run-in period, all subjects will consume provided meals. The total duration of the trial will be ~10 weeks for the older subjects, including screening, 2-wk run-in, and 6 wk of intervention, as well as ~4 weeks for the younger subjects including screening and 2-wk run-in. In addition to consuming the provided meals for 6 weeks, the older volunteers will take an assigned supplement daily. Blood samples of the older volunteers will be collected at the end of the run-in and the end of the 6-wk intervention. These same samples will only be collected from the younger volunteers at the end of the run-in period.

Older subjects will be randomly assigned to receive one of the supplements (PLA vs. FVS) after their eligibility is confirmed. A randomization scheme will be prepared by a biostatistician using a standardized computer program for two treatment groups using a parallel design.

The study supplements will be generously provided by Juice PLUS (Collierville, TN). A matching placebo product will be manufactured by the Juice PLUS under the FDA GMP guidelines. The main ingredient of the placebo will be microcrystalline cellulose-containing 0.5% magnesium stearate. The Juice PLUS products that will be used in this intervention have been marketed in the US. Microcrystalline cellulose and magnesium stearate have a GRAS status under FDA Code of Federal Regulations (CFR) title 21. FVS in a capsule form will be the combination of Juice Plus+ Garden Blend, Juice Plus+ Orchard Blend, and Juice Plus+ Berry Blend. All Juice Plus+ supplements contain a fine, granular powder, mainly from botanical ingredients. This powder is encapsulated in a size 00 gelatin capsule. These three formulas will be blended to produce a uniform brown powder and packaged into study opaque capsules.

Juice Plus+ Garden Blend consists of vegetable juice powder and pulp from carrot, parsley, beet, kale, broccoli, cabbage, spinach, oat, rice, and tomato; gelatin, glucomannan, calcium ascorbate, mixed tocopherols, calcium carbonate, garlic powder, Spirulina Pacifica, natural mixed carotenoids, natural enzyme blend, Lactobacillus acidophilus, folic acid. The powder looks pale green in color and smells like cabbage. Juice Plus+ Orchard Blend consists of fruit juice powder and pulp from apple, orange, pineapple, cranberry, peach, acerola cherry, beet, prune, date, and papaya; gelatin, calcium ascorbate, citrus pectin, citrus bioflavonoids, glucomannan, natural mixed carotenoids, natural enzyme blend, bromelain, papain, mixed tocopherols, Lactobacillus acidophilus, folic acid. The powder looks pink in color and smells like apple/cranberry. Juice Plus+ Berry Blend consists of fruit juice and pulp powder of Concord grape, blueberry, cranberry, blackberry, bilberry, raspberry, black currant, elderberry, cocoa powder, pomegranate powder, green tea, ginger root, grape seed, and artichoke leaf powder, gelatin, mixed tocopherols, calcium ascorbate, natural enzyme blend, silicon dioxide, vegetable-derived magnesium stearate, citrus bioflavonoids from tangerine, folic acid. The powder looks purple in color and smells faintly of berry and cocoa.

During the trial, older subjects will be required to attend 1 screening visit and 3 study visits over 10 weeks, and younger subjects will be required to attend 1 screening visit and 2 study visits over 4 weeks. An initial screening visit (Visit 1) is employed to obtain informed consent and determine each subject's eligibility. A blood sample will be collected only if the subject is fasting >12 hours. At Visit 2, subjects will begin to consume the provided meals for 2 weeks during the run-in period. At Visit 3, all subjects will be asked to arrive at the study site after fasting for >12 h, blood will be collected. For younger subjects, the study will complete at end of Visit 3. Older subjects will be randomly assigned to one of 2 supplements, starting on the next day of Visit 3 for 6 weeks. They will be instructed to take 3 capsules each with breakfast and dinner. At Visit 4 (final visit), older subjects will be asked to arrive at the study site after fasting for >12 h, blood will be collected for analyses.

Younger and older subjects will consume provided meals for 2 and 8 weeks. The study meals will be designed to be comparable to a diet that most average Americans are consuming. Subjects may consume the study meals longer than 2 or 8 weeks because of a visit scheduling conflict or other unexpected events.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy
2. Age, ≥55 y old
3. BMI, ≥27 and <35 kg/m2
4. Consume a typical American diet, <3 servings of combined fruits and vegetables daily
5. Waist:hip ratio >0.8 for women and >0.9 for men, and waist:height ratio ≥0.5
6. Willing to consume study meals for 8 wk
7. Do not have allergic reaction to plant foods
8. Willing to take the assigned supplement for 6 wk

Exclusion Criteria:

1. Unusual dietary pattern, including vegan/vegetarian
2. Cigarette smoking and/or nicotine replacement use in the last 6 months
3. Intend to be pregnant, pregnancy, and breastfeeding
4. Use of medications known to change lipid metabolism
5. Steroid use, except nasal and non-prescription topical treatments
6. Active treatment for cancer of any type >1 y, except non-melanoma skin cancer
7. Have an immunodeficiency condition
8. Use of immunosuppressive medications within the last 6 months
9. Weekly alcoholic intake >14 drinks (168 oz beer, 56 oz wine, 14 oz hard liquor)
10. Drugs known to influence fecal microbiota: Regular use of fiber supplements such as Metamucil, probiotics, prebiotics, laxatives, stool softeners, H2 blockers, proton pump inhibitors (PPI) or antacids.
11. Antibiotic use within 3 months prior to or during study participation
12. Colonoscopy or colonoscopy prep within 3 months prior to or during study
13. Infrequent (<3/wk) or excessive (>3/d) number of regular bowel movements
14. History of a bilateral mastectomy with nodal dissection
15. Consume ≥3 servings of fruits and vegetables daily one average
16. Gastrointestinal diseases, conditions, or medications influencing gastrointestinal absorption including active peptic ulcer disease or inflammatory bowel disease which will be found based on the self-report during the screening visit
17. Diabetes and/or use of diabetes medications
18. Unstable thyroid disease or adjustment of thyroid medication in past 6 months
19. Abnormal values of standard blood biochemistries that interfere with study outcomes based on study physician's discretion
20. Infection or immunization within 30 days prior to study admission
21. Use anticoagulants, such as heparin, warfarin (coumadin), or Plavix in past 6 months
22. On or planning to be on a weight loss regimen
23. Gain or loss of ≥5% body weight in the last 6 months
24. Inability to refrain from ASA/NSAID/Tylenol use x 720 prior to study blood draws
25. Regular use of any dietary supplements containing vitamins, minerals, herbal or other plant-based preparations, fish oil supplements (including cod liver oil) prebiotics, probiotics or homeopathic remedies; however, subjects who are willing to refrain from the use of these supplements 30 days prior to enrollment and throughout the entire study may be considered eligible

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
mitochondrial function | at end of 6-week intervention
  Targeted central carbon metabolomic in peripheral blood mononuclear cells

SECONDARY OUTCOMES:
metabolomics | at end of 6-week intervention
  non-targeting plasma metabolomics

OTHER OUTCOMES:
phytochemical concentrations in plasma | at end of 6-week intervention
  Concentrations of plasma phenolics, carotenoids, and tocopherols

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No